CLINICAL TRIAL: NCT04352816
Title: A Multi-centre Observational Cohort Trial to Identify Magnetocardiography (MCG) Parameters in the Prediction of Future ICD Therapy
Brief Title: Magnetocardiography (MCG) Parameters in the Prediction of Future ICD Therapy
Acronym: Magneto-SCD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Coventry and Warwickshire NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: FO401218
Record Dates: First submitted 2019-12-03; First posted 2020-04-20 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Death, Sudden, Cardiac; Ventricular Arrythmia
MeSH Terms: conditions — Death, Sudden, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (Experimental): Participants who do not receive an ICD therapy and have normal Echocardiogram findings and no evidence of arrhythmia will form this group. These participants will receive an MCG scan in addition to their standard care plan We will record the findings of any/all investigations participants receive as per their standard care plan, such as imaging providing left ventricular ejection fraction and usual care blood tests although their research activity/involvement in the trial will cease after the baseline observation. There will be no follow up. We aim to recruit 210 participants to this group to match the anticipated size of the group who receive an ICD but don't receive a shock.
  Interventions: Device: Magnetocardiogram
- Observation group (Experimental): The participants who go on to receive an ICD therapy, as part of standard care, will constitute the 'Observation' group. These participants will undergo an MCG, lying and standing blood pressure and undertake a quality of life questionnaire. Participants in this group will undergo additional blood tests, circulating vascular biomarkers such as (High sensitivity Troponin, Nt pro BNP, CRP, High sensitivity CRP, mRNA, IL-6). All scans and tests that are conducted as part of standard care for evaluation of requirement of ICD implantation will be collected, for example; Echocardiographic, CMRI or MUGA measurements of the heart chambers and function. We will record these findings as this will enable us to substratify patients according to different degrees of cardiac dysfunction
  Interventions: Device: Magnetocardiogram
- Device in situ group (Experimental): To achieve the secondary objectives of exploring whether features consistent with arrhythmogenesis are extractable from MCG scans on participants with ICDS and pacemakers in situ, the investigators will recruit an additional 30 participants separate from the main trial. Twenty participants will be recruited from the ICD clinic. These participants, who have already had an ICD implanted will be selected with a 50:50 split as to whether they have had previous therapy from the ICD. The presence of an ICD can impact the analysis of MCGs in these patients due to the background signal noise subtraction required to obtain a usable signal. We will use these scans to trial different signal noise reduction strategies. These will be analysed to determine whether the features seen in the main trial can be extracted from this data set.
  10 participants will be recruited who have got an upgrade from a pacemaker to an ICD.
  Interventions: Device: Magnetocardiogram

INTERVENTIONS:
Device: Magnetocardiogram — Magnetocardiography (MCG) is a non-invasive, non-contact body-surface method which uses magnetometers to measure and map the magnetic fields generated by the electrical activity within the heart. It offers a better spatial resolution than an ECG recording and opens the possibility of detecting conduction characteristics consistent with arrhythmogenesis.9-15 The application of MCG has been limited by feasibility as devices up to now have been based on superconducting quantum interference devices (SQUID) with supercooled sensors. These machines were often operated in a shielded environment, to decrease magnetic field interference (noise) from electrical devices and other sources of magnetic fields. This was a major limiting factor in deploying these devices in a working environment especially considering, that most hospital wards will have numerous devices that can interfere with the device.

SUMMARY:
A multi-centre observational cohort trial to identify Magnetocardiography (MCG) parameters in the prediction of future ICD therapy. To show a correlation between Arrhythmogenic features on MCG and future ICD therapies seen on ICD interrogation of patients at risk of SCD.

DETAILED DESCRIPTION:
AIM: To explore if VitalScan MCG parameters are able to predict future ICD therapies in patients who meet the requirements for ICD therapy.

Magnetocardiography (MCG) Magnetocardiography (MCG) is a non-invasive, non-contact body-surface method which uses magnetometers to measure and map the magnetic fields generated by the electrical activity within the heart. It offers a better spatial resolution than an ECG recording and opens the possibility of detecting conduction characteristics consistent with arrhythmogenesis.

The application of MCG has been limited by feasibility as devices up to now have been based on superconducting quantum interference devices (SQUID) with super cooled sensors. These machines were often operated in a shielded environment, to decrease magnetic field interference (noise) from electrical devices and other sources of magnetic fields. This was a major limiting factor in deploying these devices in a working environment especially considering, that most hospital wards will have numerous devices that can interfere with the device.

The investigators will be evaluating the use of a portable magnetometer which measures the change in magnetic fields rather than an absolute magnetic field as measured by SQUID magnetometers used in the trials mentioned above. It has been developed to be more affordable and more feasible than SQUID magnetometers as it is designed to be operated at room temperature in an unshielded environment. The investigators will be evaluating its ability to measure parameters identified in previous literature as well as other novel parameters that may be identified from acquiring the MCG derivative. With the development of this portable magnetometer designed to be used in an unshielded environment, there is real potential for screening a large numbers of patients for SCD risk. Until this trial, this novel tool has not been evaluated in this role.

MCG parameters in Sudden Cardiac Death (SCD) Whilst there are limited data on the role of MCG in predicting arrhythmic events, a series of studies involving patients with ischaemic heart disease have shown a correlation between MCG characteristics and the presence of ventricular arrhythmias. Specifically QRS fragmentation and late fields of the QRS have been associated with a higher incidence of ventricular arrhythmia. A trial of 49 patients with dilated cardiomyopathy demonstrated parameters present on MCG scans which were able to distinguish between participants, retrospectively, who had a ventricular arrhythmia in comparison to those who did not. The authors associated the features in the MCG T wave (specifically prolongation of the end part of the T wave) with the presence of ventricular arrhythmias. Kawakami et al prospectively studied ventricular arrhythmia risk in 51 patients with non-ischaemic cardiomyopathy for a mean follow-up of 2.9 years. They found that MCG left intraventricular disorganised conduction described as a deviation from the typical global clockwise LV depolarisation was predictive of major adverse cardiac events..

Proposed trial The aim of this trial is to show a correlation between features consistent with arrhythmogenic substrate from a VitalScan MCG and future ventricular arrhythmias; measured from observed arrhythmic events from ICD interrogation of patients at risk of SCD. The investigators hope therefore to describe MCG features most predictive of future ventricular arrhythmias.

To achieve this aim the investigators plan to perform a multi-centre cohort trial in all patients referred to cardiology at University Hospitals Coventry and Warwickshire NHS Trust and University Hospital of North Midlands. In addition to usual care, participants will have lying and standing blood pressure measured, blood samples taken for the measurement of circulating vascular biomarkers and an MCG performed. Participants will then be segregated by whether their usual treatment pathway involves or has involved the implantation of an ICD. Those patients who do not require an ICD will not receive any further follow up, but will be used to form a control group of patients. Participants who have received an ICD will be observed for any arrhythmic events for a minimum of one year.

At twelve months participants will be requested to complete a quality of life questionnaire; SF-36 to assess impact of symptoms on their quality of life. Twelve months after the recruitment of the last patient the first phase of the trial will conclude.

The second phase of the trial involves long term follow up of participants having ICD implants, for duration of five years. This will be observational and participants will not be expected to be involved in any activity above and beyond standard care.

Trial Summary The trial is a dual phase, multi-centre observational cohort trial, attempting to define the parameters of Magnetocardiography (MCG), with an aim to interpret the characteristics of these parameters, which can predict future ventricular arrhythmia and ICD therapies.

Phase one will last a total of 30 months: 12 months to recruit patients, further 18 months to complete patient follow up and for analysis of data.

If the recruitment target is not met at the 12 month time point, there will be an option to extend this period for a further 6 months.

Phase two will involve long term follow up of the cohort of participants who receive an ICD. This will allow longer time for events requiring ICD therapy to occur. This will involve an annual data collection and reporting. This will continue for five years after the recruitment of the last participant.

Study population:

The investigators plan to recruit 510 prospective participants in total out of which 300 ±10% in the observation arm (as shown in Figure 1) and 210 participants in the control arm. This will ensure sample size integrity assuming a possible 10% loss to follow up. Prospective participants will be recruited from two sites. All trial visit and procedures will be conducted in the University Hospital Coventry and Warwickshire (UHCW) and University Hospital of North Midlands (UHNM) NHS Trusts.

ELIGIBILITY:
Inclusion Criteria:

* All patients referred to the cardiology team who meet the following criteria will be invited to participate in the trial:
* Age: 18 years or over
* Can give informed consent

Exclusion Criteria:

* - Patients unable to lie still on a bed at a maximum of 30 degree angle for 5 minutes
* Patients with ongoing myocardial infarction or active ischaemia.
* Clinically unstable patients as determined by their treating clinician.
* Patients with existing thoracic metallic implants ie. pacing or defibrillator device, metallic valve will be excluded from the main arm of the trial. The research team will perform a side arm (Device in situ group) trial on 30 participants with either ICDs or pacemakers.
* Age: Under 18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2019-08-09 (Actual); Primary Completion 2021-11-17 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with features of heterogenous myocardial conduction (eg. late QRS signals, QT dispersion) and correlation with ventricular arrhythmias as reported by ICD interrogation | 12-72 months
  We will remotely follow up participants who have had ICD and observe if they have had an ICD interrogation (Shock) for arrythmogenic events. These are defined by ventricular rates that are faster than 149 beats per minute and deemed to be ventricular in origin on ICD interrogation during standard follow up. We will the compare the MCG scans of participants who had shock with that of whom did not.

SECONDARY OUTCOMES:
Exploring the correlation of MCG QRS fragmentation and current flow analysis with ICD therapies | 12-72 months
  Outcome measures - ICD therapies: ICD interrogation (Shock) for arrythmogenic events. These are defined by ventricular rates that are faster than 149 beats per minute and deemed to be ventricular in origin on ICD interrogation during standard follow up.
  MCG: QRS fragmentation as defined by waveform extrema and amplitude in normalised MCG waveform.
  Current flow analysis is derived from MCG field maps and is perpendicular to the magnetic field.
Exploring the correlation between ECG parameters, Echo findings, MCG parameters and ICD therapies. | 12-72 months
  Outcome measures - ICD therapies: ICD interrogation (Shock) for arrythmogenic events. These are defined by ventricular rates that are faster than 149 beats per minute and deemed to be ventricular in origin on ICD interrogation during standard follow up.
  ECG parameters: QRS width
  Echo parameters: Left Ventricular Ejection Fraction - categorised into participants with severely impaired systolic function (LVEF<35%) or those without (LVEF>35%)
  MCG parameters: Features of heterogenous conduction (eg. late QRS signals, QT dispersion)
Correlation of MCG parameters with Left ventricular ejection fraction (LVEF) | Baseline
  LVEF as determined by Echo or CMRI expressed as % change in LV volume during cardiac cycle
  MCG parameters: Features of heterogenous conduction (eg. late QRS signals, QT dispersion)
Analysis of the SF-36 quality of life questionnaire results | 12 month follow up
  Evaluate the responses to a SF-36 quality of life questionnaire to document the tolerability of ICD implantation and therapy.
  Comparisons will be made between responses from those participants who have received therapy from their device and those who haven't and between those participants who have a primary or secondary indication for their device.

CONTACTS AND LOCATIONS:
Overall Officials: Faizel Osman, MD FRCP FESC, Principal Investigator — university Hospital Coventry and Warwickshire
Locations (1):
- University Hospital Coventry and Warwickshire NHS Trust, Coventry, West Midlands, United Kingdom

REFERENCES:
- [Derived] Lachlan T, He H, Sharma K, Khan J, Rajappan K, Morley-Davies A, Patwala A, Randeva H, Osman F. MAGNETO cardiography parameters to predict future Sudden Cardiac Death (MAGNETO-SCD) or ventricular events from implantable cardioverter defibrillators: study protocol, design and rationale. BMJ Open. 2020 Oct 10;10(10):e038804. doi: 10.1136/bmjopen-2020-038804. PMID 33040013